CLINICAL TRIAL: NCT03116971
Title: A Multicenter Study With an Open Label Phase Ib Part Followed by a Randomized, Placebo-controlled, Double-blind, Phase II Part to Evaluate Efficacy, Safety, Tolerability, and PK of M3814 in Combination With Etoposide and Cisplatin in Subjects With Treatment-naïve Small Cell Lung Cancer (SCLC) Extensive Disease (ED)
Brief Title: Phase Ib/II Study of M3814 With Etoposide and Cisplatin in Small Cell Lung Cancer (SCLC) Extensive Disease (ED)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment in the study was prematurely terminated due to recruitment challenges and not due to concerns of safety for the participants.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS100036-0022
Record Dates: First submitted 2017-03-28; First posted 2017-04-17 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Small Cell Lung Cancer
Keywords: M3814, Small Cell Lung Cancer (SCLC), Deoxyribonucleic acid-dependent protein kinase inhibitor, Chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — peposertib; Cisplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- M3814 PiC with Etoposide and Cisplatin (Experimental): Participants received M3814 100 milligram (mg) powder in capsule (PiC) orally once daily in combination with Etoposide 100 mg/m^2 over a 60 minute intravenous infusion on Days 1-3 and Cisplatin 75 milligram per square meter (mg/m^2) over a 60-minute intravenous infusion on Day 1 for 6 cycles with each cycle lasting 3 weeks (21 days) until progressive disease (PD).
  Interventions: Drug: M3814; Drug: Cisplatin; Drug: Etoposide
- M3814 (HME Tablet + PiC) with Etoposide and Cisplatin (Experimental): Participants received M3814 100 mg hot melt extrusion (HME) tablet orally 5 days prior to Day 1 and M3814 100 mg PiC, orally once daily from Day 1 in combination with Etoposide 100 mg/m^2 over a 60 minute intravenous infusion on Days 1-3 and Cisplatin 75 mg/m^2 over a 60-minute intravenous infusion on Day 1 for 6 cycles with each cycle lasting 3 weeks (21 days) until PD.
  Interventions: Drug: M3814; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: M3814 — Participants received M3814 PiC or hot melt extrusion (HME) tablet orally once daily in combination with etoposide (intravenously) and cisplatin for 6 cycles with each cycle lasting 3 weeks (21 days).
  Other Names: MSC2490484A; Peposertib
Drug: Cisplatin — Cisplatin 75 milligram per square meter (mg/m^2) was administered over a 60-minute intravenous infusion on Day 1.
Drug: Etoposide — Etoposide 100 mg/m^2 over a 60 minute IV infusion on Days 1-3 was administered for 6 cycles with each cycle lasting 3 weeks (21 days).

SUMMARY:
M3814 is an investigational drug under evaluation for treatment of lung cancer. The purpose of the study was to assess the Safety and Efficacy of M3814 in combination with chemotherapy with SCLC ED.

DETAILED DESCRIPTION:
The study was intended to be a phase I/II trial, but the study never moved forward to Phase II due to recruitment challenges.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study (Phase Ib and Phase II) the participant must fulfill all of the following criteria:

* Male or female participants at least 18 years of age
* Histological or cytological diagnosis of SCLC
* Extensive disease (ie, disease beyond ipsilateral hemithorax, which may include malignant pleural or pericardial effusion or hematogenous metastases [Tany, Nany, M1a/b; T3-T4, Nany, M0, due to multiple lung nodules or extent of disease that precludes a tolerable radiation field, as judged by the Investigator])
* Participants eligible for first line platinum-based chemotherapy
* Measurable or evaluable disease according to RECIST v1.1
* Eastern Cooperative Oncology Group performance status (ECOG PS) less than equals to (<=) 2
* Life expectancy of greater than equals to (≥) 3 months
* Female participants of childbearing potential and male participants with female partners of childbearing potential must be willing to avoid pregnancy Note: Other protocol defined criteria could apply.

Exclusion Criteria:

Participants are not eligible for the study if they fulfill any of the following exclusion criteria:

* Prior anticancer therapy for extensive disease (ED) SCLC including experimental agents.
* Concurrent use of other anticancer therapy including any investigational agent within 28 days prior to the first dose of the investigational drug M3814.
* Extensive prior radiotherapy (RT) on more than 30% of bone marrow reserves (by Investigator judgment)
* Prior bone marrow/stem cell transplantation within 5 years before study start (Phase II only)
* Major surgical intervention within 28 days prior to the first dose of investigational drug administration. Intervention(s) to establish the diagnosis for SCLC is permitted within 28 days as long as participants are cleared by the medical and surgical teams.
* Poor vital organ functions defined as:
* Bone marrow impairment as evidenced by hemoglobin less than (<) 9.0 gram per deci liter (g/dL) (5.7 micromole per liter (μmol/L)), absolute neutrophil count < 1.5 × 109/L, platelets < 100 × 109/L
* Renal impairment as evidenced by calculated creatinine clearance < 60 mL/minutes (min) (according to the Cockcroft-Gault formula)
* Liver function abnormality as defined by total bilirubin greater than (>) 1.5 × upper limit of normal (ULN) or aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5 × ULN (participants with liver involvement: a maximum of AST/ALT 5 × ULN)
* Contraindication to the use of etoposide or cisplatin
* Participants currently receiving (or unable to stop using prior to receiving the first dose of investigational drug) medications or herbal supplements known to be potent inhibitors of cytochrome P450 (CYP) 3A and CYP2C19 (unless treatment can be discontinued at least 1 week prior to receiving the first dose of investigational drug) or potent inducers of CYP3A and CYP2C19 (unless treatment can be discontinued at least 3 weeks prior to receiving the first dose of investigational drug). Note: Other protocol defined criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Number of Subjects Experienced Any Dose-Limiting Toxicity (DLT) over the DLT period. | up to 21 days
Phase Ib: Determination of Recommended Phase II dose (RP2D) of Escalating Dose of M3814 in Combination With Cisplatin and Etoposide for the Phase II Part of the Study | up to 11 months
Phase II: Progression Free Survival (PFS) as Assessed by the Investigator according to RECIST v1.1 | Time from randomization to first assessment of disease progression or death, whichever is earlier, assessed up to 24 months
  PFS time will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause.

SECONDARY OUTCOMES:
Phase Ib: Number of Subjects with of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Deaths | From the first dose of study drug treatment up to 30 days after the last dose of study drug treatment
  An Adverse Event (AE) is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Phase Ib: Number of Subjects with Abnormal Laboratory Values, Abnormal Vital Signs and Abnormal Electrocardiograms (ECGs) | From the first dose of study drug treatment up to 30 days after the last dose of study drug treatment
  Subjects will be analyzed for vital signs (eg, body temperature, respiratory rate, heart rate, and blood pressure), laboratory parameters and 12-lead ECG recorded at baseline and after administration of M3814. Number of subjects with abnormal values for laboratory values, vital signs and electrocardiograms (ECGs) will be reported.
Phase Ib: Change in Eastern Cooperative Oncology Group performance status (ECOG PS) | From the first dose of study drug treatment up to 30 days after the last dose of study drug treatment
Phase Ib: Percentage of Subjects with Objective Response (OR) According to RECIST v1.1 | Post randomization with period tumor evaluations until disease progression or subject withdrawal of consent, irrespective of treatment discontinuation or initiation of another therapy, assessed up to 11 months
  The Objective Response Rate (ORR) is defined as the percentage of subjects whose Best objective response (BOR) is either complete response (CR) or partial response (PR). The ORR will be derived from the BOR according to response evaluation criteria in solid tumors (RECIST) v1.1 as assessed by the Investigator.
Phase Ib: Duration of Response (DoR) According to RECIST v1.1 | First documented complete response or partial response, whichever is first recorded until the first assessment of disease progression, assessed up to 11 months
  The DoR applies only to subjects whose BOR is either CR or PR. The duration is measured from the first documented response (CR or PR, whichever is first recorded) until the first assessment of Progressive Disease (PD).The DoR will be derived from the BOR according to RECIST v1.1 as assessed by the Investigator.
Phase Ib: Percentage of Subjects With Disease Control | First documented complete response or partial response, whichever is first recorded until the first assessment of disease progression, assessed up to 11 months
  Percentage of subjects with disease control as assessed by best overall response of either CR, PR or Stable Disease (SD) will be reported.
Phase Ib: Progression Free Survival (PFS) According to RECIST v1.1 | Time from randomization to first assessment of disease progression or death, whichever is earlier, assessed up to 11 months
  The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause. The PFS will be derived according to RECIST v1.1 as assessed by the Investigator.
Phase Ib: Overall Survival (OS) | Time from randomization to death due to any cause, assessed up to 11 months
  The OS time is defined as the date from randomization to death due to any cause.
Phase Ib: Area under the concentration-time curve from 0 to 4 hours (AUC 0-4), 0 to 24 hours (AUC 0-24) for M3814, Cisplatin and Etoposide | Day (D) -1, Cycle (C) 1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hours (hrs) post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose, C3D1 Pre-dose and 3.5 hrs post dose
Phase Ib: Area Under the Concentration-Time Curve From Time 0 to the Last Quantifiable Concentration (AUC 0-t ) for M3814, Cisplatin and Etoposide | Day (D) -1, Cycle (C) 1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase Ib: Maximum Observed Plasma Concentration (Cmax) for M3814, Cisplatin and Etoposide | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post-dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post-dose, C2D3 Pre-dose
Phase Ib: Time to Reach Maximum Plasma Concentration (Tmax) for M3814, Cisplatin and Etoposide | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post-dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post-dose, C2D3 Pre-dose
Phase Ib: Apparent Terminal Half-life (t1/2) for M3814 | C1D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hours (hrs) post-dose
Phase Ib: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of M3814 | C1D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hours (hrs) post-dose
Phase Ib: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of M3814 | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post-dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post-dose, C2D3 Pre-dose
Phase Ib: Intravenous (IV) Clearance (CL) of Cisplatin and Etoposide | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hr post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase Ib: Apparent Volume of Distribution Following Extravascular Administration (Vz/f) of M3814 | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase Ib: Apparent Volume of Distribution (Vz) of Cisplatin and Etoposide | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase Ib: Terminal rate constant (λz) for M3814, Cisplatin and Etoposide | Day (D) -1, C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase Ib: Changes in Cmax for M3814 Between Day -1 and C2D1 | Day (D) -1, Cycle (C) 2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose
Phase Ib: Changes in AUC for M3814 Between Day -1 and C2D1 | Day (D) -1, Cycle (C) 2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose
Phase Ib: Changes in AUC for Etoposide From C1D1 to C1D2, C1D3, and C2D1 (for the first 2 dose levels), or From C1D1 to C2D1 (other dose levels) | Day (D) -1, Cycle (C) 1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose
Phase Ib: Changes in Cmax for Etoposide From C1D1 and C2D1 | Cycle (C) 1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose
Phase Ib: Changes in AUC for Cisplatin From C1D1 to C1D2, C1D3, and C2D1 (for the first 2 dose levels), or From C1D1 to C2D1 (other dose levels) | Day (D) -1, Cycle (C) 1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose
Phase Ib: Changes in Cmax for Cisplatin From C1D1 and C2D1 | Cycle (C) 1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5 (excluding D-1), 4, 6 and 8 hours (hrs) post dose
Phase II: Overall Survival (OS) | Time from randomization to death due to any cause, assessed up to 24 months
Phase II: Percentage of Subjects with Objective Response (OR) According to RECIST v1.1 | Post randomization every 6 weeks up to Week 54 and then every 12 weeks until disease progression or subject withdrawal of consent, irrespective of treatment discontinuation or initiation of another therapy., assessed up to 24 months
  The Objective Response Rate (ORR) is defined as the proportion of subjects whose Best objective response (BOR) is either complete response (CR) or partial response (PR). The ORR will be derived from the BOR according to response evaluation criteria in solid tumors (RECIST) Version 1.1 as assessed by the Investigator.
Phase II: Duration of Response (DoR) According to RECIST v1.1 | First documented complete response or partial response, whichever is first recorded until the first assessment of disease progression, assessed up to 24 months
  The DoR applies only to subjects whose BOR is either CR or PR. The duration is measured from the first documented response (CR or PR, whichever is first recorded) until the first assessment of Progressive Disease (PD).The DoR will be derived from the BOR according to RECIST v1.1 as assessed by the Investigator.
Phase II: Percentage of Subjects With Disease Control | First documented complete response or partial response, whichever is first recorded until the first assessment of disease progression, assessed up to 24 months
  Percentage of subjects with disease control as assessed by best overall response of either CR, PR or Stable Disease (SD) will be reported.
Phase II: Percentage of Subjects Who Received Prophylactic Cranial Irradiation (PCI) and/or Thorax Irradiation After 6 Cycles of Treatment | After 6 Cycles of treatment, assessed up to 24 months
Phase II: Tumor shrinkage From Baseline in target lesions | Post randomization every 6 weeks up to Week 54 and then every 12 weeks until disease progression or subject withdrawal of consent, irrespective of treatment discontinuation or initiation of another therapy., assessed up to 24 months
Phase II: Number of subjects with of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Deaths | From the first dose of study drug treatment up to 30 days after the last dose of study drug treatment
  An Adverse Event (AE) is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious AE (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Phase II: Number of Subjects with Abnormal Laboratory Values, Abnormal Vital Signs and Abnormal Electrocardiograms (ECGs) | From the first dose of study drug treatment up to 30 days after the last dose of study drug treatment
Phase II: Change in Eastern Cooperative Oncology Group performance status (ECOG PS) | From the first dose of study drug treatment up to 30 days after the last dose of study drug treatment
Phase II: Primary Health-Related Quality of Life (HRQoL) Based on Time to Definitive Deterioration (TUDD) as Assessed Using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | Screening; Post randomization every 6 weeks up to Week 54 and then every 12 weeks until disease progression or subject withdrawal of consent, irrespective of treatment discontinuation or initiation of another therapy., assessed up to 24 months
Phase II: Primary HRQoL based on TUDD Assessed Using EORTC Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) | Screening; Post randomization every 6 weeks up to Week 54 and then every 12 weeks until disease progression or subject withdrawal of consent, irrespective of treatment discontinuation or initiation of another therapy., assessed up to 24 months
Phase II: Primary HRQoL based on TUDD Assessed Using European Quality of Life 5- dimensions questionnaire (EQ-5D) | Screening; Post randomization every 6 weeks up to Week 54 and then every 12 weeks until disease progression or subject withdrawal of consent, irrespective of treatment discontinuation or initiation of another therapy., assessed up to 24 months
Phase II: Area under the concentration-time curve from 0 to 24 hours (AUC 0-24) for M3814, Cisplatin and Etoposide | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC 0-t ) for M3814, Cisplatin and Etoposide | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Maximum Observed Plasma Concentration (Cmax) for M3814, Cisplatin and Etoposide | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Time to Reach Maximum Plasma Concentration (Tmax) for M3814, Cisplatin and Etoposide | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Apparent Terminal Half-life (t1/2) for M3814 | C1D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose
Phase II: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of M3814 | C1D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose
Phase II: Total Body Clearance From Plasma Following Extravascular Administration (CL/f) of M3814 | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Intravenous (IV) Clearance (CL) of Cisplatin and Etoposide | Time Frame: C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Apparent Volume of Distribution Following Extravascular Administration (Vz/f) of M3814 | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose
Phase II: Apparent Volume of Distribution (Vz) of Cisplatin and Etoposide | C1D1, C2D1: Pre-dose, 0.5, 1, 1.5, 2, 3, 3.5, 4, 6 and 8 hrs post dose; C1D2 Pre-dose, C1D3 Pre-dose, C1D8 Pre-dose, C1D15 Pre-dose and 2 hrs post dose, C2D3 Pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (79):
- United States (16):
  - Research site, Mesa, Arizona
  - Research site 1, Santa Rosa, California
  - Research site, Santa Rosa, California
  - Research site, Whittier, California
  - Research site, Danbury, Connecticut
  - Research site, Norwalk, Connecticut
  - Research site, Columbus, Georgia
  - Research site, Newnan, Georgia
  - Research site, Topeka, Kansas
  - Research site, Ashland, Kentucky
  - Research site, Billings, Montana
  - Research site, Pinehurst, North Carolina
  - Research site, Cincinnati, Ohio
  - Research site, Portland, Oregon
  - Research site, Philadelphia, Pennsylvania
  - Research site, Houston, Texas
- Belgium (8):
  - Research site, Aalst
  - Research site, Charleroi
  - Research site, Edegem
  - Research site, Ghent
  - Research site, Libramont
  - Research site, Liège
  - Research site, Roeselare
  - Research site, Yvoir
- Bulgaria (6):
  - Research site 4, Sofia
  - Research site 2, Sofia
  - Research site 6, Sofia
  - Reasearch site 5, Sofia
  - Research site 3, Sofia
  - Research site 1, Sofia
- Canada (4):
  - Research site, Calgary, Alberta
  - Research site, Saint John, New Brunswick
  - Research site, London, Ontario
  - Research site, Toronto, Ontario
- Czechia (2):
  - Research site, Benešov
  - Research site, Olomouc
- Denmark (3):
  - Research site, Aalborg
  - Research site, Herlev
  - Research site, Odense C
- Germany (9):
  - Research site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research site, Gauting, Bavaria
  - Research site, Nuremberg, Bavaria
  - Research site, Hanover, Lower Saxony
  - Research site, Chemnitz, Saxony
  - Research site, Kiel, Schleswig-Holstein
  - Research site, Lübeck, Schleswig-Holstein
  - Research site 1, Berlin
  - Research site 2, Berlin
- Hungary (6):
  - Research site 1, Budapest
  - Research site 2, Budapest
  - Research site 3, Budapest
  - Research site, Farkasgyepű
  - Research site, Szekszárd
  - Research site, Szolnok
- Italy (8):
  - Research site, Rozzano, Milano
  - Research site, Catania
  - Research site, Genova
  - Research site, Napoli
  - Research site, Ravenna
  - Research site, Reggio Emilia
  - Research site, Roma
  - Research site, Torino
- Poland (4):
  - Research site, Olsztyn
  - Research site, Poznan
  - Research site, Warsaw
  - Research site, Wodzisław Śląski
- Romania (4):
  - Research site, Baia Mare
  - Research site, Cluj-Napoca
  - Research site, Craiova
  - Research site, Timișoara
- Spain (5):
  - Research site, Badajoz
  - Research site 1, Madrid
  - Research site 4, Madrid
  - Research site 3, Madrid
  - Research site 2, Madrid
- United Kingdom (4):
  - Research site, Hull, East Riding Of Yorkshire
  - Research site, London, Greater London
  - Research site, Sheffield, South Yorkshire
  - Research site, Glasgow, Strathclyde